CLINICAL TRIAL: NCT03281148
Title: Evaluation of Accuracy in Computer Guided Versus Free Hand Immediate Implant Placement in Fresh Extraction Sockets: a Randomized Controlled Clinical Trial
Brief Title: Accuracy in Computer Guided Versus Free Hand Immediate Implantation
Acronym: RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Mohammed Ayman, Assistant lecturer at Prosthodontic Department Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Prosthetic department
Record Dates: First submitted 2017-09-10; First posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Immediate Dental Implants
Keywords: immediate implants, accuracy,extraction sockets

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer guided implant insertion group (Experimental): According to the allocation, the experimental group will receive implants immediately placed in extraction sockets using CAD/CAM surgical guides.
  Interventions: Device: Computer guided implant insertion group
- Free hand implant insertion group (Active Comparator): According to the allocation, the control group will receive implants immediately placed in extraction sockets using traditional free hand technique.
  Interventions: Device: Free hand implant insertion group

INTERVENTIONS:
Device: Computer guided implant insertion group — Implants will be immediately inserted in fresh extraction sockets using CAD/CAM guides
  Arms: Computer guided implant insertion group
Device: Free hand implant insertion group — Implants will be immediately inserted in fresh extraction sockets using free hand technique
  Arms: Free hand implant insertion group

SUMMARY:
Patients with hopeless teeth in the esthetic area requiring immediate implant restoration will be recruited to the study. Patients will be divided into two groups; a group will receive immediate implants placed using CAD/CAM guides while the other group will receive immediate implants placed by free hand technique. Accuracy of inserted implants will be measured.

DETAILED DESCRIPTION:
Interventions The principal investigator (DA) will diagnose all patients and select them according to inclusion and exclusion criteria.

The principal investigator (DA) will prepare all patients. Patient preparation will take few steps that are important for optimum planning of implant insertion and restoration. Actual treatment steps will start after preparation is done including; surgical and prosthetic procedures.

1. Case history

   1. Medical history:

      The principal investigator (DA) will ask all patients about their present and previous systemic condition and any history of hospitalization or surgeries. Controlled diabetic patients will be asked to bring a recent blood glucose test. This includes both fasting/post prandial &glycosylated hemoglobin test (Hemoglobin A1c) to evaluate their current status.
   2. Dental history:

      The principal investigator (DA) will ask all patients about past dental procedures including implants.

      b) Clinical examination

   <!-- -->

   1. Visual examination:

      The principal investigator (DA) will examine all patients extra orally to assess the temporomandibular joints, temporalis, and masseter muscle to help in detection of bruxism. Intraoral examination includes assessment of any pathological lesion (cyst/tumor) that may interfere with the planned implant treatment.
   2. Digital examination:

      The principal investigator (DA) will examine the soft tissue surrounding hopeless teeth digitally using index finger to confirm a firm mucosa free from any flabby tissue, absence of severe undercuts and absence of abnormal ridge contour. The principal investigator (DA) will examine the bone volume arbitrary using the two index fingers to confirm an adequate bucco-lingual bone width. The principal investigator (DA) will test tooth mobility of adjacent teeth using a periodontal probe to ensure that the remaining adjacent teeth are not mobile.

      c) Construction of scan appliance: The principal investigator (DA) will make primary upper and lower impressions for the selected patients using irreversible hydrocolloid impression material in stock trays of suitable sizes. The principal investigator (DA) will pour impressions using Type IV extra hard dental stone . The principal investigator (DA) will take a Face bow record and a diagnostic bite record for each patient using Utility Wax . A semi-adjustable articulator will be used for mounting.

      A diagnostic mock up for broken/ badly decayed teeth will be formed for needed patients. By pressing a clear thermoplastic sheet using a vacuum forming machine on the study cast of the patient; a vacuum formed template will be constructed containing radiopaque markers for easy superimposition later. The vacuum template is now considered the scan appliance.

      d) Patient Radiographic Imaging Every patient will be then sent for a CBCT scanning for the upper and/or lower arch. The patient will be instructed to wear the scan appliance during imaging. Midline will be adjusted using laser beam and a scout will be taken to the patient. The patient will be asked to stay still till the machine rotates around him/her. The cone beam computed tomography images will be obtained in Digital Imaging & Communications in Medicine (DICOM) format on a compact disc.

      e) Virtual planning and construction of surgical guide

      a) Virtual Planning The CBCT image was used for the virtual surgical and prosthetic planning of implant placement using Blusky® software. First, the remaining and neighboring teeth will be segmented. This step helped in virtually inserting implants in an acceptable position in relation to neighboring teeth with respect to their crowns and roots. Virtual Setting will be done then virtual insertion of implants with appropriate sizes will be done with respect to the future prosthesis.

      Cautious respect to anatomical landmarks in the area of interest will be considered during planning. In the mandible; Mandibular canal will be simulated to be seen in both 2D and 3D views. In the maxilla; maxillary sinus lining will be checked in all views during implant positioning.

      A Virtual guide will be designed from the CBCT of the patient to be seated on neighboring teeth. The exported Standard Language transformation (STL) file of the virtual guide will be sent to labs centers by e-mail for construction.

      f) Surgical Procedures: The Principal investigator (DA) will extract the remaining root or tooth in an atraumatic procedure procedure using lancet, periotome, minimal force and rotational movement. After extraction the socket will be examined for intact labial and palatal bone using depth probe. If all walls are intact the socket would be eligible for immediate implant placement.

      In the test group, the computer guided surgical guide will be used for implant drilling and placement following the manufacturer's instructions.

      While in the control group, after tooth or root extraction implants will be placed free hand guided by the extraction sockets.

      Then in implants with primary stability (Insertion torque> 35 Ncm2), the final abutment will be placed and any further adjustment would be done immediately in the lab and re-positioned in place. The principal investigator (DA) will check the vacuum stent is in its place again intraorally, then a chair side tooth colored auto-polymerizing resin will be injected into the vacuum sheet corresponding to the implant site to construct the temporary crown.

      If any subject is to feel any movement in his/her temporary crown, an immediate phone call is to be done to (DA) to examine the cause of mobility (whether it is the crown only or the implant itself).

      g) Postoperative Care: The principal investigator (DA) will manage postoperative complications. The principal investigator (DA) will remove mobile temporary crowns and recement them. While mobile implants will be considered as early stage failed implants and it will be removed immediately. The patient will receive another implant at the same site after a proper healing period of at least 3 months during which he/she will be provided with a temporary removable partial denture for aesthetics.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hopeless teeth or remaining roots
2. Bucco-lingual bone thickness of 7mm or more (Spray et al., 2000)
3. Bucco-lingual keratinized mucosa of 6mm or more (Spray et al., 2000)
4. Inter-arch space sufficient for prosthetic rehabilitation (7mm or more) (Misch, 2008)
5. Adults more than 18 years old

Exclusion Criteria:

1. Uncontrolled diabetic patients (HbA1c value ≥ 8.1 percent) (Takeshita et al., 1998)(Javed & Romanos, 2009)(Garg, 2010)(Retzepi & Donos, 2010)(B R Chrcanovic et al., 2014)
2. Heavy smokers (More than 10 cigarettes per day) (Nitzan et al., 2005) (Strietzel et al., 2007) (Abt, 2009)(Bruno Ramos Chrcanovic et al., 2015)
3. Severe bruxers (Lobbezoo et al., 2006) (Manfredini et al., 2011)(Lin et al., 2012)(Zhou et al., 2015)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Linear Deviation | two months postoperative
  The amount of linear deviation was measured through three parameters; global, lateral and depth deviation. These parameters will be measured at the apical and coronal center in a mesiodistal and buccolingual plane.

CONTACTS AND LOCATIONS:
Overall Officials: Maha ElKerdawy, Professor, Study Chair — Professor at Faculty of Dentistry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alzoubi, Fawaz, Nima Massoomi, and A. N. (2016). Accuracy Assessment of Immediate and Delayed Implant Placements Using CAD/CAM Surgical Guides. Journal of Oral Implantology ., 42(5), 391-398. http://doi.org/10.1002/smll.)) D'haese, J., Van De Velde, T., Komiyama, A., Hultin, M., & De Bruyn, H. (2012). Accuracy and complications using computer-designed stereolithographic surgical guides for oral rehabilitation by means of dental implants: a review of the literature. Clinical Implant Dentistry and Related Research, 14(3), 321-35. http://doi.org/10.1111/j.1708-8208.2010.00275.x Ortega-martínez, J., Pérez-pascual, T., Mareque-bueno, S., & Hernández-alfaro, F. (2012). Immediate implants following tooth extraction . A systematic review. Medicina Oral Patología Oral Y Cirugia Bucal- Oral Surgery Section, 17(2), e251-61. http://doi.org/10.4317/medoral.17469